CLINICAL TRIAL: NCT07069114
Title: Impact of Prognostic Factors on Treatment Outcomes in Patients With Cervical Degenerative Disc Disease Undergoing Anterior Cervical Discectomy and Fusion With the Bagby and Kuslich (BAK/C) Technique: A Retrospective Cohort Study
Brief Title: Prognostic Factors for ACDF With BAK/C in Cervical Disc Disease
Status: Completed | Type: Observational
Sponsor: Liang Hao (Other)
Responsible Party: Sponsor-Investigator, Liang Hao, Principal Investigator, The Third Hospital of Shijiazhuang
Organization: The Third Hospital of Shijiazhuang (Other)
Other Study IDs: 2023-B056
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Favorable Outcome Group (Control Group): Patients (n=52) who underwent ACDF with BAK/C and achieved good neurological recovery, defined as Visual Analog Scale (VAS) ≤ 2 combined with a Japanese Orthopaedic Association (JOA) score improvement of ≥4 points at 3-year follow-up.
  Interventions: Procedure: Anterior Cervical Discectomy and Fusion with BAK/C Interbody Fusion
- Poor Outcome Group (Observation Group): Patients (n=28) who underwent ACDF with BAK/C and demonstrated minimal or worsened neurological recovery, defined as VAS > 2 with a JOA improvement of <2 points or neurological deterioration at 3-year follow-up.
  Interventions: Procedure: Anterior Cervical Discectomy and Fusion with BAK/C Interbody Fusion

INTERVENTIONS:
Procedure: Anterior Cervical Discectomy and Fusion with BAK/C Interbody Fusion — The surgical intervention consisted of anterior cervical discectomy and fusion (ACDF). Patients were placed under general anesthesia in a supine position with slight neck extension. A standard right anterior cervical approach was utilized to expose the affected vertebral levels. Following the removal of the degenerated intervertebral disc and osteophytes, the interbody space was prepared. A Bagby and Kuslich (BAK/C) interbody fusion cage, filled with autogenous bone fragments, was implanted to facilitate fusion. In cases of multi-level surgery, an anterior cervical plate was selectively applied for enhanced stability based on intraoperative assessment. Postoperatively, all patients were required to wear a Philadelphia hard neck brace for a period of 2 months.

SUMMARY:
This retrospective study aimed to identify predictive prognostic factors for treatment outcomes in patients with cervical degenerative disc disease (CDDD). The study analyzed data from 80 patients who underwent anterior cervical discectomy and fusion (ACDF) with the Bagby and Kuslich (BAK/C) technique. Patients were stratified into two groups based on clinical outcomes at a 3-year follow-up, and logistic regression was used to determine which factors, such as age and bone mineral density, were independent predictors of poor recovery.

DETAILED DESCRIPTION:
Cervical degenerative disc disease (CDDD) is a prevalent condition causing significant pain and neurological dysfunction. Anterior cervical discectomy and fusion (ACDF) combined with the Bagby and Kuslich (BAK/C) interbody fusion technique is an established surgical treatment, but patient outcomes vary. This study was designed to address a gap in the literature by retrospectively analyzing both surgical and patient-related variables over a 3-year follow-up period to understand the factors influencing treatment success. A cohort of 80 patients treated between January and December 2020 was identified. Patients were divided into a "favorable outcome" group and a "poor outcome" group based on post-operative pain relief and neurological improvement (JOA score). The study's primary objective was to use multivariate logistic regression analysis to identify independent risk factors (e.g., age, bone mineral density, disease severity, postoperative complications) associated with poor outcomes. The findings aim to provide evidence-based insights to help optimize patient selection and treatment strategies for ACDF with BAK/C fusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18, regardless of gender.
* Diagnosed with degenerative cervical intervertebral disc disease based on clinical and imaging findings.
* Significant pain and symptoms impacting quality of life, requiring surgery.
* Undergoing anterior decompression and BAK/C interbody fusion.
* Minimum 3-year follow-up data available.

Exclusion Criteria:

* Serious cervical conditions (e.g., fracture, infection, tumor).
* Previous cervical surgery or other treatments.
* Pregnant or lactating women.

Ages: 36 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hospitalized patients diagnosed with symptomatic cervical degenerative disc disease who were treated at The Third Hospital of Shijiazhuang. The cohort was derived from a consecutive series of patients who underwent anterior cervical discectomy and fusion (ACDF) with the BAK/C technique between January and December 2020. The final included sample of 80 patients had a mean age of 55.36 years (range 36-75) and were selected based on specific inclusion/exclusion criteria, including the absence of prior cervical surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of Independent Risk Factors for Poor Surgical Outcomes | Assessed based on data collected up to the 3-year final follow-up
  To identify predictors of poor treatment outcome using multivariate logistic regression analysis. The analysis evaluated variables including age, bone mineral density, baseline disease severity (initial JOA score), postoperative complications, and postoperative care. The outcome was being classified into the "Poor Outcome Group".

SECONDARY OUTCOMES:
Change in Neurological Function | Baseline (preoperative), 1 week postoperative, 6 months postoperative, and 3-year final follow-up
  Assessed using the Japanese Orthopaedic Association (JOA) scoring system, which ranges from 0 (severe impairment) to 17 (normal function).
Radiological Fusion Rate | Assessed at 6 months and at the 3-year final follow-up
  Assessed via X-ray and CT scans. Firm fusion was defined as segmental motion <2 degrees on extension-flexion radiographs and bridging trabecular bone across ≥50% of the graft-host interface. The rate of pseudoarthrosis (non-fusion) was reported as a key radiological outcome.
Change in Intervertebral Height | 1 week postoperative and 3-year final follow-up
  Measured from lateral X-ray images. The change was calculated as the difference between the immediate postoperative height and the height at the final follow-up.
Incidence of Postoperative Complications | Assessed throughout the 3-year follow-up period
  Number and type of adverse events recorded, including C5 palsy and pseudoarthrosis, categorized as intraoperative, early postoperative (<30 days), or late postoperative (>30 days).
Bone Mineral Density (BMD) | Baseline (Preoperative)
  Measured preoperatively using dual-energy X-ray absorptiometry (DXA) at the lumbar spine and reported as a T-score to assess bone quality.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Shijiazhuang, Shijiazhuang, Hebei, China